CLINICAL TRIAL: NCT04924699
Title: A Study of MRG002 in the Treatment of Patients With HER2-positive Unresectable Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-004
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Breast Cancer (BC)
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRG002 (Experimental): MRG002 will be administrated via intravenous infusion of 2.6 mg/kg once on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002
- Trastuzumab Emtansine for Injection (Active Comparator): Trastuzumab Emtansine for Injection will be administrated via intravenous infusion of 3.6 mg/kg once on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: Trastuzumab Emtansine for Injection

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously
  Arms: MRG002
Drug: Trastuzumab Emtansine for Injection — Administrated intravenously
  Arms: Trastuzumab Emtansine for Injection

SUMMARY:
The primary objective of Phase II is to evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of MRG002 in patients with HER2-positive, unresectable locally advanced or metastatic breast cancer. The primary objective of Phase III is to evaluate the efficacy and safety of MRG002 versus Trastuzumab Emtansine (T-DM1) in patients with HER2-positive unresectable locally advanced or metastatic breast cancer who have been previously treated with trastuzumab (or a biosimilar) and an anti-HER2 tyrosine kinase inhibitor (anti-HER2-TKI) and have progressed on or after the most recent therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 to 75 (including 18 and 75)，both genders;

  2. Expected survival time ≥ 6 months;

  3. The score of ECOG for performance status is 0 or 1;

  4. Patients with histologically and/or cytologically confirmed HER2-positive invasive breast cancer, including unresectable locally advanced breast cancer (LABC) or metastatic breast cancer (MBC);

  5. Phase II: patients with advanced or metastatic disease who have previously failed trastuzumab (containing trastuzumab biosimilar) ± pertuzumab and taxane, or progressed within 12 months after neoadjuvant or adjuvant therapy (using trastuzumab (containing trastuzumab biosimilar) ± pertuzumab and taxane regimen); patients who have failed TKI and/or HER2-targeted ADCs can also be included. Phase III: patients who have received 1 or 2 prior lines of anti-HER2 therapy for locally advanced or recurrent/metastatic breast cancer (in the case of (neo) adjuvant therapy, such (neo) adjuvant therapy also counts as one line of anti-HER2 therapy if relapse occurs within 12 months of (neo) adjuvant therapy); have received prior treatment with trastuzumab (containing a trastuzumab biosimilar) and anti-HER2-TKI; have not received prior treatment with ADCs;

  6. Patients must have imaging evidence of tumor progression during or after the most recent treatment confirmed by the investigator and have at least one measurable lesion baseline according to RECIST 1.1;

  7. Organ functions must meet the basic requirements;

  8. Reproductive male and female patients of childbearing age shall be willing to take effective contraceptive measures from the date of signing the ICF to 6 months after the last dose. Women of childbearing potential must have a negative pregnancy test within 7 days before the first dose.

Exclusion Criteria:

* 1. History of other primary malignancies;

  2. Received investigational drugs from other clinical trials, any anti-tumor drugs, or radiotherapy within 4 weeks prior to the first dose/randomization; or use of endocrine therapy for breast cancer within 7 days prior to the first dose/randomization, or have current requirement of endocrine therapy; or have received strong CYP3A4 inhibitors or inducers within 2 weeks prior to the first dose/randomization, or have current requirement of CYP3A4 inhibitors or inducers; cumulative doxorubicin up to 450 mg/m2 or equivalent prior to the first dose/randomization; or had major surgery within 4 weeks prior to the first dose/randomization without full recovery or planned surgery within 12 weeks after study treatment;

  3. Presence of central nervous system (CNS) metastasis;

  4. The pleural or peritoneal effusion with combined clinical symptoms, which seriously endangers the life safety of the subjects or urgently needs clinical treatment. Or the pericardial effusion with combined clinical symptoms;

  5. Any severe or uncontrolled systemic disease, uncontrolled heart disease, uncontrolled diabetes, and active bleeding signs judged by the investigator;

  6. Evidence of active infection, including hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection, active bacteria infection requiring systematic anti-infective therapy, infection caused by other viruses, fungi, rickettsia or parasites;

  7. History of hypersensitivity to any component of MRG002 or history of hypersensitivity of ≥ Grade 3 to trastuzumab injection;

  8. Subjects with active autoimmune disease or a history of autoimmune disease are receiving immunosuppressive agents or systemic hormone therapy, and are still receiving within 2 weeks prior to enrollment/randomization;

  9. History of interstitial pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc;

  10. Other conditions inappropriate for participation in this study, as deemed by the investigator;

  11. Presence of peripheral neuropathy > Grade 1;

  12. History of cirrhosis (decompensated cirrhosis Child-Pugh class B, C).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by Independent Review Committee (IRC) | Baseline to study completion（up to 36 months）
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause assessed by Independent Review Committee (IRC) according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion (up to 36 months)
  ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) according to RECIST v1.1.
Duration of Response (DoR) | Baseline to study completion (up to 36 months)
  DoR is defined as the time from first documented objective response (CR/PR) to the first onset of tumor progression or death of any nonsurgical cause.
Disease Control Rate (DCR) | Baseline to study completion (up to 36 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and stable disease (SD) after treatment.
PFS by investigator | Baseline to study completion (up to 36 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 36 months)
  OS is defined as the duration from the start of treatment to death of any cause.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Concentration-time curve | Baseline to 30 days after the last dose of study treatment
  Plot of drug concentration changing with time after drug administration.
Immunogenicity | Baseline to 30 days after the last dose of study treatment
  The proportion of patients with positive ADA immunogenicity results.

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, Doctor, Principal Investigator — Fifth Medical Center of PLA General Hospital; Yunjinang Liu, Doctor, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (19):
- China (19):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Fourth hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hosipital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shengyang, Liaoning
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing, Tianjing
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No